CLINICAL TRIAL: NCT05859867
Title: Bimbingamba Zerosix Third Phase: Studying Communities
Acronym: Bimbingamba
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliero Universitaria Maggiore della Carita (Other)
Collaborators: Compagnia di San Paolo (Other)
Responsible Party: Principal Investigator, Flavia Prodam, Associated Prof. in Clinical Nutrition and MD, Azienda Ospedaliero Universitaria Maggiore della Carita
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CE273/2022
Record Dates: First submitted 2023-04-12; First posted 2023-05-16 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Obesity; Childhood Obesity; Weight Loss; Life Style, Healthy
Keywords: Childhood Obesity
MeSH Terms: conditions — Obesity; Pediatric Obesity; Weight Loss | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Children resident in the Municipality of Mondovì (Intervention group) (Experimental): Recruiting of 1000 children (more or less) with ages between 0 and 5 years resident in the Municipality of Mondovì.
  Eligible subjects are children with a date of birth between 1/1/2018 and 31/12/2022 (subjects born in 5 years prior to the start of the project), plus a cohort of newborn between 01/1/2023 and 21/6/2023.
  Children of both sex and of any ethnicity could be enrolled in the trial.
  Moreover, parents of eligible and enrolled children are also considered in-study subjects.
  Interventions: Other: Promotion of Healthy Nutrition and Physical Activity
- Children resident in the Municipality of Savigliano (Control group) (No Intervention): Recruiting of 1000 children (more or less) with ages between 0 and 5 years resident in the Municipality of Savigliano.
  Eligible subjects are children with a date of birth between 1/1/2018 and 31/12/2022 (subjects born in 5 years prior to the start of the project), plus a cohort of newborn between 01/1/2023 and 21/6/2023.
  Children of both sex and of any ethnicity could be enrolled in the trial.
  Moreover, parents of eligible and enrolled children are also considered in-study subjects.

INTERVENTIONS:
Other: Promotion of Healthy Nutrition and Physical Activity — Through scheduled and specific activities, enrolled subjects receive information for the promotion of the Mediterranean diet and Mediterranean lifestyle habits, according to the pyramid of the Mediterranean diet. In addition, subjects receive general recommendations about the promotion of regular recreational motor activity, the pyramid of physical activity for pediatric age, and free games appropriate to age. These activities are conducted by professionals in the food (nutritionists) and sports sectors and are aimed in the preparation of simple recipes repeatable at home, and in motor play activities to encourage physical activity. Information regarding clinical, and socio-demographic parameters and family habits will be collected through validated questionnaires.
  Arms: Children resident in the Municipality of Mondovì (Intervention group)

SUMMARY:
Childhood obesity is increasing in the last years especially in developed countries, and, as well as adult obesity, is related to the development of pathologies. Unfortunately, the restoration of a normal weight condition, if the ponderal excess rose in the first years of life, seems very difficult. Despite the importance of this issue, there is a paucity of evidence demonstrating effective interventions in reducing weight over time. The observation that in developed countries childhood obesity appears with evident social and geographical gradients justifies the implementation of inter-sectoral interventions of primary prevention, to be declined at the contextual level: family and community. Nowadays, there are numerous interventions for the promotion of lifestyle in pediatric age, in particular, those aimed at primary school and adolescence. On the other hand, few interventions were directed at the 0-7 age group.

Therefore, this community intervention trial involved the pediatric population (aged 0-7 years) and their families, and it is aimed at the prevention of obesity and the restoring normal weight through community interventions aimed at improving lifestyles and with them the bio-metric parameters, health and well-being outcomes and soft skills in the population aged 0-7 years.

The target population is children aged 0-7 years resident in the two municipalities (Mondovì and Savigliano), respectively selected as Intervention and Control Common. Totally, to conduct this study 2000 children, of both sex, will be enrolled (near 1000 for each of the two Municipalities).

DETAILED DESCRIPTION:
Bimbingamba is an initiative promoted by "Fondazione Compagnia di San Paolo" with the aim of achieving healthy nutrition and physical exercise among children, aged 0-7 years. The initiative will take place in Mondovì (Cuneo, Italy), selected as the intervention Municipality, and will involve resident children with their families. Due to the common interest in the topic, Compagnia di San Paolo has requested the University of Eastern Piedmont of collaborating on the project.

As reported by literature, childhood obesity presents a multifactorial origin being determined by the interaction between environmental and genetic factors. Increased habits in consuming "junk foods", sweetened beverages, unhealthy lifestyles, and low levels of physical activity are the major driving factors for the development of obesity during childhood. The restoration of a normal weight condition, especially if the ponderal excess rose in the first years of life, seems very difficult to achieve not only because of behavioral mechanisms but also of epigenetic imprinting. The interest of this study is the prevention of the obese phenotype in children together with the restoration of normal weight. There are a great number of interventions centered on the promotion of a healthy lifestyle in adolescents, but few of these are focused on infancy, especially interventions directed to the 0-7 age group. According to reported knowledge, preventing obesity in childhood is important for reducing the risk of obesity among adolescents and adults. Therefore preventing/reducing the related comorbidities.

This intervention study will be conducted in two Italian Commons, Mondovì and Savigliano, respectively selected as the interventional Municipality and control Municipality. The study will include at least 200 children between 0-7 years with their families living and residing in one of the two cities. The main objectives of this study will be the description of weight status during the time in the 0-7 aged group in relation to the socio-economic factors, parental parameters, families, and lifestyle habits. As a secondary objective, this study aims to evaluate the effectiveness of interdisciplinary interventions in the community. Therefore, evaluating lifestyle promotion, health improvement, and soft skills acquisition in the 0-7 aged group.

Interventions will be administered during organized events involving the participation of children and their families together with the presence of specialized staff (nutritionists, personal trainers, educators). During these days children will be educated in the Mediterranean diet and healthy cooking (preparing simple meals with their parents) guided by nutritionists and will be involved in recreational and motor activities to promote physical activity.

Participants' recruiting will occur during the organized events, in places of birth, kindergarten, and vaccination centers through informative materials. On the occasion of the first meeting, those parents apparently interested will be given the materials and the link for the application (https://bimbingambazerosei.app.interacta.space/) through which join the projects and fill out the informed consent for them and their children. Recruiting period will start in April 2023.

Data collection will be performed by the specialized personnel by using specific and validated questionnaires, by taking clinical and non-clinical data, and by data arriving from health sources (i.e.: emergency accesses). All data will be registered in REDCap.

The study is thought to last 2 years, pre-intervention data will be collected at time (t) 0 (during recruiting), while post-intervention data will be collected at t24 (end of the study). Among the possible outcomes of treatment have been identified the percentage of children that are average weight or overweight, the number of children having a Mediterranean diet regimen before and after the educational period, the kind of family diet, and the level of physical activity.

Obtained data will be analyzed with statistical analysis (i.e. ANOVA and t.test) in order to identify the differences between the intervention and the control group. The final aim of the study is to obtain different data among the two cohorts regarding the prevalence of risk factors related to obesity, among the adherence of children and their families to the Mediterranean diet, differences in anthropometric and clinical parameters, and the ability of parents in distinguish healthy and unhealthy habits for their children.

The entire study will be conducted according to the Helsinki Declaration and following the Standards of Good Clinical Practice of the European Union.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 0-5 year of both sex resident in the two Municipalities under evaluation
* children having date of birth between 1/1/2018 and 31/12/2022 (subjects born 5 years prior to the start of the project)
* newborns between 01/1/2023 and 21/6/2023 residing in the two municipalities under study.

Exclusion Criteria:

* Residence/domicile in the municipalities under investigation, for a period of time less than 6 months following recruitment;
* Recruitment of the child in other intervention trials of any nature.

Ages: 2 Days to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 2000 (Estimated)
Dates: Start 2023-04-15 (Actual); Primary Completion 2025-04-15 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of weigh/overweight subjects | Change in body weight at time 0 and 24 months.
  Variation in total body weight in children belonging to the intervention or control groups at times 0 and 24 months.
Rate of Mediterranean Diet (MD) adherence | Change in KIDMED score at time 0 and 24 months.
  Variation in nutritional habits (Western Diet to Mediterranean Diet) in both control and intervention groups at times 0 and 24 months. Habits in consuming MD are evaluated with KIDMED (Mediterranean Diet Quality Index) questionnaire, the scores are as follows:
  total score = 12 points lower than 3 = low adherence to MD between 4-7= moderate adherence to MD higher than 8= high adherence to MD
Physical activity level | Change in IPAQ score at time 0 and 24 months.
  Variation in physical activity level assessed by the International Physical Activity Questionnaire "IPAQ" in both control and intervention groups at time t0 and 24 months.
  IPAQ scale is based on MET (minutes of physical activity per week):
  lower than 30 minutes per day = low level of physical activity equal to 30 minutes per day= moderate level of physical activity higher than 3000 minutes per week (MET)= high level of physical activity
Adherence to Mediterranean Diet | Changes in the adherence of Mediterranean Diet between 0 and 24 months.
  Evaluate the Mediterranean Diet adherence (consumption of fruit, vegetables, nuts, extra virgin olive "EVO" oil, and so on) before and after the intervention in both control and intervention groups.
  The questionnaire will be performed on time t0 (time of enrollment) and time t24 (24 months later).
  This questionnaire gives as results the percentage of macronutrient and micronutrient consumption and the association with Mediterranean Diet adherence.
Nutritional habits | Changes in nutritional habits between time 0 and 24 months
  Nutritional habits will be evaluated in both the control and intervention groups through the use of the Andromeda questionnaire. This questionnaire will be performed at time 0 (during the enrollment) and 24 months later.
  Andromeda is a questionnaire that collects information on eating habits in terms of the frequency of food consumption in the last year. Therefore, the questionnaire assesses dietary habits before the start of the observation period (t0) and 24 months (two years) after the observation or intervention period.
  There is no score for this questionnaire, it divides food into macro-categories giving information about the nutrients assumption.
Access rate to Emergency Room (ER) and Pediatricians of Free Choice (PFC) | Changes in the ER and PFC accesses at time 0 and 24 months.
  Comparison in number of times visiting ER and PFC among the intervention and control group at times 0 and 24 months.
Change in physiological parameters | Variation in Likert scale points at time 0 and 24 months.
  Variation in self-confidence, self-control, and socialization level in control and intervention groups at times 0 and 24 months. These physiological parameters are evaluated through the use of Likert scale having 5 points:
  1. Very satisfied.
  2. Moderately satisfied.
  3. Neither satisfied nor dissatisfied.
  4. Moderately dissatisfied.
  5. Very dissatisfied

CONTACTS AND LOCATIONS:
Locations (1):
- University of Eastern Piedmont, Novara, Italy

REFERENCES:
- [Background] Archero F, Ricotti R, Solito A, Carrera D, Civello F, Di Bella R, Bellone S, Prodam F. Adherence to the Mediterranean Diet among School Children and Adolescents Living in Northern Italy and Unhealthy Food Behaviors Associated to Overweight. Nutrients. 2018 Sep 18;10(9):1322. doi: 10.3390/nu10091322. PMID 30231531
- [Background] Belot M, James J. Healthy school meals and educational outcomes. J Health Econ. 2011 May;30(3):489-504. doi: 10.1016/j.jhealeco.2011.02.003. Epub 2011 Mar 1. PMID 21458872
- [Background] Colquitt JL, Loveman E, O'Malley C, Azevedo LB, Mead E, Al-Khudairy L, Ells LJ, Metzendorf MI, Rees K. Diet, physical activity, and behavioural interventions for the treatment of overweight or obesity in preschool children up to the age of 6 years. Cochrane Database Syst Rev. 2016 Mar 10;3(3):CD012105. doi: 10.1002/14651858.CD012105. PMID 26961576
- [Background] Craig CL, Marshall AL, Sjostrom M, Bauman AE, Booth ML, Ainsworth BE, Pratt M, Ekelund U, Yngve A, Sallis JF, Oja P. International physical activity questionnaire: 12-country reliability and validity. Med Sci Sports Exerc. 2003 Aug;35(8):1381-95. doi: 10.1249/01.MSS.0000078924.61453.FB. PMID 12900694
- [Background] Crispim SP, Nicolas G, Casagrande C, Knaze V, Illner AK, Huybrechts I, Slimani N. Quality assurance of the international computerised 24 h dietary recall method (EPIC-Soft). Br J Nutr. 2014 Feb;111(3):506-15. doi: 10.1017/S0007114513002766. Epub 2013 Sep 4. PMID 24001201
- [Background] Davison KK, Gavarkovs A, McBride B, Kotelchuck M, Levy R, Taveras EM. Engaging Fathers in Early Obesity Prevention During the First 1,000 Days: Policy, Systems, and Environmental Change Strategies. Obesity (Silver Spring). 2019 Apr;27(4):525-533. doi: 10.1002/oby.22395. PMID 30900405
- [Background] Di Cesare M, Soric M, Bovet P, Miranda JJ, Bhutta Z, Stevens GA, Laxmaiah A, Kengne AP, Bentham J. The epidemiological burden of obesity in childhood: a worldwide epidemic requiring urgent action. BMC Med. 2019 Nov 25;17(1):212. doi: 10.1186/s12916-019-1449-8. PMID 31760948
- [Background] Estruch R, Ros E, Salas-Salvado J, Covas MI, Corella D, Aros F, Gomez-Gracia E, Ruiz-Gutierrez V, Fiol M, Lapetra J, Lamuela-Raventos RM, Serra-Majem L, Pinto X, Basora J, Munoz MA, Sorli JV, Martinez JA, Fito M, Gea A, Hernan MA, Martinez-Gonzalez MA; PREDIMED Study Investigators. Primary Prevention of Cardiovascular Disease with a Mediterranean Diet Supplemented with Extra-Virgin Olive Oil or Nuts. N Engl J Med. 2018 Jun 21;378(25):e34. doi: 10.1056/NEJMoa1800389. Epub 2018 Jun 13. PMID 29897866
- [Background] Ferrari P, Kaaks R, Fahey MT, Slimani N, Day NE, Pera G, Boshuizen HC, Roddam A, Boeing H, Nagel G, Thiebaut A, Orfanos P, Krogh V, Braaten T, Riboli E; European Prospective Investigation into Cancer and Nutrition study. Within- and between-cohort variation in measured macronutrient intakes, taking account of measurement errors, in the European Prospective Investigation into Cancer and Nutrition study. Am J Epidemiol. 2004 Oct 15;160(8):814-22. doi: 10.1093/aje/kwh280. PMID 15466504
- [Background] Giordano L, Gallo F, Petracci E, Chiorino G, Segnan N; Andromeda working group. The ANDROMEDA prospective cohort study: predictive value of combined criteria to tailor breast cancer screening and new opportunities from circulating markers: study protocol. BMC Cancer. 2017 Nov 22;17(1):785. doi: 10.1186/s12885-017-3784-5. PMID 29166878
- [Background] Gonzalez CA. The European Prospective Investigation into Cancer and Nutrition (EPIC). Public Health Nutr. 2006 Feb;9(1A):124-6. doi: 10.1079/phn2005934. PMID 16512959
- [Background] Vineis P, Riboli E. The EPIC study: an update. Recent Results Cancer Res. 2009;181:63-70. doi: 10.1007/978-3-540-69297-3_7. No abstract available. PMID 19213558
- [Background] Hennessy M, Heary C, Laws R, van Rhoon L, Toomey E, Wolstenholme H, Byrne M. The effectiveness of health professional-delivered interventions during the first 1000 days to prevent overweight/obesity in children: A systematic review. Obes Rev. 2019 Dec;20(12):1691-1707. doi: 10.1111/obr.12924. Epub 2019 Sep 2. PMID 31478333
- [Background] Larque E, Labayen I, Flodmark CE, Lissau I, Czernin S, Moreno LA, Pietrobelli A, Widhalm K. From conception to infancy - early risk factors for childhood obesity. Nat Rev Endocrinol. 2019 Aug;15(8):456-478. doi: 10.1038/s41574-019-0219-1. Epub 2019 Jul 3. PMID 31270440
- [Background] Liu Z, Xu HM, Wen LM, Peng YZ, Lin LZ, Zhou S, Li WH, Wang HJ. A systematic review and meta-analysis of the overall effects of school-based obesity prevention interventions and effect differences by intervention components. Int J Behav Nutr Phys Act. 2019 Oct 29;16(1):95. doi: 10.1186/s12966-019-0848-8. PMID 31665040
- [Background] Martinez-Gonzalez MA, Corella D, Salas-Salvado J, Ros E, Covas MI, Fiol M, Warnberg J, Aros F, Ruiz-Gutierrez V, Lamuela-Raventos RM, Lapetra J, Munoz MA, Martinez JA, Saez G, Serra-Majem L, Pinto X, Mitjavila MT, Tur JA, Portillo MP, Estruch R; PREDIMED Study Investigators. Cohort profile: design and methods of the PREDIMED study. Int J Epidemiol. 2012 Apr;41(2):377-85. doi: 10.1093/ije/dyq250. Epub 2010 Dec 20. No abstract available. PMID 21172932
- [Background] Mazarello Paes V, Ong KK, Lakshman R. Factors influencing obesogenic dietary intake in young children (0-6 years): systematic review of qualitative evidence. BMJ Open. 2015 Sep 16;5(9):e007396. doi: 10.1136/bmjopen-2014-007396. PMID 26377503
- [Background] Prina S, Royer H. The importance of parental knowledge: evidence from weight report cards in Mexico. J Health Econ. 2014 Sep;37:232-47. doi: 10.1016/j.jhealeco.2014.07.001. Epub 2014 Jul 22. PMID 25132149
- [Background] Reilly JJ, Martin A, Hughes AR. Early-Life Obesity Prevention: Critique of Intervention Trials During the First One Thousand Days. Curr Obes Rep. 2017 Jun;6(2):127-133. doi: 10.1007/s13679-017-0255-x. PMID 28434107
- [Background] Reinehr T. Long-term effects of adolescent obesity: time to act. Nat Rev Endocrinol. 2018 Mar;14(3):183-188. doi: 10.1038/nrendo.2017.147. Epub 2017 Nov 24. PMID 29170543
- [Background] Serra-Majem L, Ribas L, Ngo J, Ortega RM, Garcia A, Perez-Rodrigo C, Aranceta J. Food, youth and the Mediterranean diet in Spain. Development of KIDMED, Mediterranean Diet Quality Index in children and adolescents. Public Health Nutr. 2004 Oct;7(7):931-5. doi: 10.1079/phn2004556. PMID 15482620
- [Background] Strauss RS. Childhood obesity and self-esteem. Pediatrics. 2000 Jan;105(1):e15. doi: 10.1542/peds.105.1.e15. PMID 10617752
- [Background] Valerio G, Maffeis C, Saggese G, Ambruzzi MA, Balsamo A, Bellone S, Bergamini M, Bernasconi S, Bona G, Calcaterra V, Canali T, Caroli M, Chiarelli F, Corciulo N, Crino A, Di Bonito P, Di Pietrantonio V, Di Pietro M, Di Sessa A, Diamanti A, Doria M, Fintini D, Franceschi R, Franzese A, Giussani M, Grugni G, Iafusco D, Iughetti L, Lamborghini A, Licenziati MR, Limauro R, Maltoni G, Manco M, Reggiani LM, Marcovecchio L, Marsciani A, Del Giudice EM, Morandi A, Morino G, Moro B, Nobili V, Perrone L, Picca M, Pietrobelli A, Privitera F, Purromuto S, Ragusa L, Ricotti R, Santamaria F, Sartori C, Stilli S, Street ME, Tanas R, Trifiro G, Umano GR, Vania A, Verduci E, Zito E. Diagnosis, treatment and prevention of pediatric obesity: consensus position statement of the Italian Society for Pediatric Endocrinology and Diabetology and the Italian Society of Pediatrics. Ital J Pediatr. 2018 Jul 31;44(1):88. doi: 10.1186/s13052-018-0525-6. PMID 30064525
- [Background] Venturelli F, Ferrari F, Broccoli S, Bonvicini L, Mancuso P, Bargellini A, Giorgi Rossi P. The effect of Public Health/Pediatric Obesity interventions on socioeconomic inequalities in childhood obesity: A scoping review. Obes Rev. 2019 Dec;20(12):1720-1739. doi: 10.1111/obr.12931. Epub 2019 Aug 29. PMID 31468647
- [Background] Muros J. J. and E. Knox (2020), Mediterranean diet and mental well-being in the young, The Mediterranean Diet. An Evidence-Based Approach, 2nd Edition - July 4, 2020, • Editors: Victor Preedy, Ronald Watson. Paperback ISBN: 9780128186497
- [Background] Blanchflower, D.G., Oswald, A.J. & Stewart-Brown, S. Is Psychological Well-Being Linked to the Consumption of Fruit and Vegetables?. Soc Indic Res 114, 785-801 (2013). https://doi.org/10.1007/s11205-012-0173-y
- [Background] Cuadros-Meñaca A., Thomsen M. R., Nayga R. M. (2022), The effect of breakfast after the bell on student academic achievement, Economics of Education Review, Volume 86, 2022.